CLINICAL TRIAL: NCT02387437
Title: Evaluation of Different Effects of Three Recruitment Maneuvers on the Lung Heterogeneity of Acute Respiratory Distress Syndrome
Brief Title: Different Effects of Three Recruitment Maneuvers on the Lung Heterogeneity of Acute Respiratory Distress Syndrome
Acronym: DEOTRMOARDS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Southeast University, China (Other)
Collaborators: Zhongda Hospital (Other)
Responsible Party: Principal Investigator, Jianfeng Xie, Director, Southeast University, China
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2014ZDSYLL124.1
Record Dates: First submitted 2015-02-04; First posted 2015-03-13 (Estimated); Last update posted 2015-03-13 (Estimated); Status verified 2014-12

CONDITIONS: Acute Respiratory Distress Syndrome
Keywords: ARDS; EIT; recruitment maneuvers
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- SI recruitment (Experimental): Compare the effect of three recruitment maneuvers before and after recruitment maneuvers is implemented,SI continuous positive airway pressure (CPAP) held at 40 cm H2O for 40 secs.
  Interventions: Behavioral: SI recruitment; Behavioral: IP recruitment; Behavioral: PCV recruitment
- IP recruitment (Experimental): Compare the effect of three recruitment maneuvers before and after recruitment maneuvers is implemented,Incremental positive end-expiratory pressure (PEEP) with a fixed peak pressure (IP), PEEP increased in 5 cm H2O increments (allowing 30 secs/step) from a baseline PEEP of post-trial to 40 cm H2O while decreasing tidal volume to limit peak inspiratory pressure to 40 cm H2O. After CPAP of 40 cm H2O was held for 30 secs, PEEP was decremented in 5-cm H2O steps to the post-RM PEEP setting, while increasing tidal volume toward the baseline value of 10 mL/kg (as the 40 cm H2O peak pressure limit allowed).
  Interventions: Behavioral: SI recruitment; Behavioral: IP recruitment; Behavioral: PCV recruitment
- PCV recruitment (Experimental): Compare the effect of three recruitment maneuvers before and after recruitment maneuvers is implemented,PCV peak pressure = 40 cm H2O, inspiratory to expiratory ratio = 1:2, and PEEP level = 15cm H2O for 2 min
  Interventions: Behavioral: SI recruitment; Behavioral: IP recruitment; Behavioral: PCV recruitment

INTERVENTIONS:
Behavioral: SI recruitment — SI continuous positive airway pressure (CPAP) held at 40 cm H2O for 40 secs.
Behavioral: IP recruitment — Incremental positive end-expiratory pressure (PEEP) with a fixed peak pressure (IP), PEEP increased in 5 cm H2O increments (allowing 30 secs/step) from a baseline PEEP of post-trial to 40 cm H2O while decreasing tidal volume to limit peak inspiratory pressure to 40 cm H2O. After CPAP of 40 cm H2O was held for 30 secs, PEEP was decremented in 5-cm H2O steps to the post-RM PEEP setting, while increasing tidal volume toward the baseline value of 10 mL/kg (as the 40 cm H2O peak pressure limit allowed).
Behavioral: PCV recruitment — PCV peak pressure = 40 cm H2O, inspiratory to expiratory ratio = 1:2, and PEEP level = 15cm H2O for 2 min

SUMMARY:
Acute respiratory distress syndrome (ARDS) is the common disease in clinical, which pathophysiology is a lot of alveolar collapse and heterogeneity. Recruitment maneuver is one of the important therapy for improvement of this phenomenon. The previous research focuses on the hemodynamic and oxygenation effect of recruitment maneuver on the lung of ARDS. Seldom investigators try to find the intuitive change of heterogeneity when recruitment maneuver is implemented. In this study, the investigators compare three recruitment maneuvers on the lung heterogeneity of ARDS.

DETAILED DESCRIPTION:
Acute respiratory distress syndrome (ARDS) is the common disease in clinical,which pathophysiology is a lot of alveolar collapse and heterogeneity. Recruitment maneuver is one of the important therapy for improvement of this phenomenon. The previous research focuses on the hemodynamic and oxygenation effect of recruitment maneuver on the lung of ARDS. Seldom investigators try to find the intuitive change of heterogeneity when recruitment maneuver is implemented. In this study, the investigators compare three recruitment maneuvers on the lung heterogeneity of ARDS.

Electrical impedance tomography (EIT) has been introduced as a true bedside and radiation-free technique which provides information on heterogeneity. The investigators compare effects of three recruitment maneuvers on lung heterogeneity before recruitment maneuver and do the same thing after three recruitment maneuvers.

Ninety-three patients with ARDS will be enrolled . These patients are treated routinly.They need to recept a time of ZEEP (PEEP is zero cmH2O)for ten respiratory cycles before RM(recruitment maneuvers).Implemente a kind of RM at random immediately after ZEEP,Then make the ventilator same as before ZEEP.The EIT images ,blood gases and hemodynamic variables will be examined as beseline between ZEEP and RM.Completion of this kind of RM lies that the P/F of blood gases 3 minutes after RM achieves (1) PO2/FiO2>400mmHg or (2)PO2/FiO2+PCO2 ≥ 400mmHg(FiO2=1)，(3)the difference between this index before lung recriument and after lung recriument PO2/FiO2<5%.In addition,3 minutes after RM,compare the indexs above between three methods.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are severe or moderate ARDS
* Patients who have signed ICF

Exclusion Criteria:

* Patients who are younger than 18 years old or older than 75 years old
* Patients whose vital signs are unstable
* Patients who are in other clinical trails
* Patients who are pregnant

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Estimated)
Dates: Start 2014-11; Primary Completion 2016-01 (Estimated); Study Completion 2016-01 (Estimated)

PRIMARY OUTCOMES:
oxygenation (improvement of oxygenation) | improvement of oxygenation 3 minutes after lung recruiment
  detection of index 3 minutes after lung recruiment (1) PO2/FiO2>400mmHg or (2)PO2/FiO2+PCO2 ≥ 400mmHg(FiO2=1)，(3)the difference between this index before lung recriument and after lung recriument PO2/FiO2<5%

CONTACTS AND LOCATIONS:
Overall Officials: Yingzi Huang, Study Director — southeast univerity, China
Locations (1):
- Zhongda hospital, Southeast University, Nanjing, Jiangsu, China